CLINICAL TRIAL: NCT05007652
Title: A Clinical Trial of KRN125 to Mobilize Hematopoietic Stem Cells Into Peripheral Blood in Patients With Multiple Myeloma and Malignant Lymphoma
Brief Title: A Study of KRN125 in Patients With Multiple Myeloma and Malignant Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125-102
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma and Malignant Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multiple myeloma cohort (KRN125) (Experimental)
  Interventions: Drug: KRN125(pegfilgrastim), PLR001(plerixafor)
- multiple myeloma cohort (KRN8601) (Active Comparator)
  Interventions: Drug: KRN8601(filgrastim), PLR001(plerixafor)
- malignant lymphoma cohort (Experimental)
  Interventions: Drug: KRN125(pegfilgrastim), PLR001(plerixafor)

INTERVENTIONS:
Drug: KRN125(pegfilgrastim), PLR001(plerixafor) — 7.2 mg of KRN125 in Day 1 Single subcutaneous administration The concomitant drug PLR001 is administered subcutaneously once daily at a dose of 0.24 mg/kg when meets the criteria. The dosing period is 12-9 hours before apheresis on the following day.
  Arms: malignant lymphoma cohort; multiple myeloma cohort (KRN125)
Drug: KRN8601(filgrastim), PLR001(plerixafor) — 400 ug/m2 of KRN8601 from Day 1 to the end date of the Apheresis Once daily subcutaneous administration The concomitant drug PLR001 is administered subcutaneously once daily at a dose of 0.24 mg/kg when meets the criteria. The dosing period is 12-9 hours before apheresis on the following day.
  Arms: multiple myeloma cohort (KRN8601)

SUMMARY:
To determine if KRN125 is non-inferior to filgrastim for the mobilization of hematopoietic stem cells into the peripheral blood in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

Criteria for the multiple myeloma cohort

* Patients with histologically or pathologically diagnosed multiple myeloma
* Patients who achieved CR, sCR, VGPR, and PR with induction therapy Criteria for the malignant lymphoma cohort
* Patients with histologically or pathologically diagnosed malignant lymphoma
* First or second CR or PR Multiple myeloma cohort, malignant lymphoma cohort common criteria
* Patients aged 20 to 75 years or younger at the time of informed consent

Exclusion Criteria:

* Those who received allogeneic hematopoietic stem cell transplantation (Allo-SCT), autologous hematopoietic stem cell transplantation (ASCT), or CAR-T therapy
* Patients who have developed adverse events leading to discontinuation of hematopoietic stem-cell collection due to administration of granulocyte colony-stimulating factor (G-CSF) or apheresis
* Patients who have not been able to collect adequate amounts of hematopoietic stem cells with G-CSF or plerixafor administration
* Patients with hypersensitivity to G-CSF or plerixafor
* Patients with ECOG Performance status (PSs) of 2 or greater.
* Patients whose cardiac or pulmonary conditions were judged to be inappropriate for apheresis or ASCT.
* Pregnant or breastfeeding female patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Achievement of a target of ≥ 2*10^6 CD34+ cells/kg collected during apheresis period in patients with multiple myeloma. | Day 5, 6, 7

SECONDARY OUTCOMES:
Achievement of a target of ≥ 2*10^6 CD34+ cells/kg collected during apheresis period in patients with malignant lymphoma. | Day 1, 4, 5, 6, 7

OTHER OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Day 30 or initiation of radiotherapy or chemotherapy
Serum KRN125 concentrations | Day 30 or initiation of radiotherapy or chemotherapy
Anti-KRN125 antibody | Day 30 or initiation of radiotherapy or chemotherapy

CONTACTS AND LOCATIONS:
Locations (21):
- Japan (21):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - The Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Hokkaido University Hospital of the National University Corporation, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - Kochi Health Sciences Center, Kochi
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Niigata University Medical and Dental Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka International Cencer Institute, Osaka
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goto H, Sawa M, Fujiwara SI, Ri M, Ishida T, Takeuchi M, Ishitsuka K, Toyosaki M, Sunami K, Tsukada J, Sonoki T, Shimogomi A, Ichihashi Y, Ouchi Y, Miyamoto T, Hino M, Maeda Y, Teshima T. Impact of single dose of pegfilgrastim on peripheral blood stem cell harvest in patients with multiple myeloma or malignant lymphoma. Sci Rep. 2025 Apr 25;15(1):14523. doi: 10.1038/s41598-025-98453-7. PMID 40281003